CLINICAL TRIAL: NCT01352468
Title: Development of a Multi-faceted Cognitive Training Program for Children With ADHD
Brief Title: Development of a Multi-faceted Cognitive Training Program for Children With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R33MH085842 (NIH); R21MH085842 (NIH)
Record Dates: First submitted 2011-03-24; First posted 2011-05-12 (Estimated); Results first posted 2017-08-01 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-06

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; cognitive training
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multifaceted Cognitive Training (Experimental): Cognitive Training with 4 different tasks each of which gets progressively more difficult as children obtain proficiency.
  Interventions: Other: Multifaceted cognitive training
- Sham Cognitive Training (Sham Comparator): Cognitive Training with 4 different tasks which does not get progressively more difficult throughout training
  Interventions: Other: Multifaceted cognitive training

INTERVENTIONS:
Other: Multifaceted cognitive training — Four computerized training tasks

SUMMARY:
After decades of Attention Deficit Hyperactivity Disorder (ADHD) intervention research, only two intervention approaches (i.e., psychopharmacology, behavioral treatment) have a "well-established" evidence-base supporting their efficacy for children with ADHD. Both of these interventions have inherent limitations. Recently multiple studies have demonstrated that cognitive training may improve neuropsychological and behavioral functioning in children with ADHD. The magnitude of treatment effects for cognitive training has been comparable to treatment effects for behavioral treatment for ADHD (i.e., small to moderate effect sizes). A limitation of existing cognitive training programs that may limit their efficacy is that each has employed a unifaceted approach. Each intervention program has targeted a single cognitive domain (e.g., working memory). This is problematic since as a group, children with ADHD have multiple areas of cognitive deficit (i.e., working memory, attention, response inhibition, delay aversion, intra-individual variability) and thus a unifaceted intervention does not address the multifaceted array of cognitive dysfunction in children with ADHD. Also, because individuals with ADHD each have unique patterns of cognitive deficits, a unifaceted cognitive training approach may target areas which are non-deficient and miss areas of significant deficit in individual patients depending on their ideographic cognitive profile. The primary goal of the proposed research is to develop and test a multifaceted cognitive training intervention that addresses a comprehensive array of ADHD-related cognitive deficits thereby ensuring that children's unique areas of cognitive deficit are targeted. During Phase I (R21 grant), software and a manual will be developed consisting of four training tasks targeting response inhibition, verbal working memory, attention, and delay aversion. Each task will possess advancing levels of difficulty. On each task, children will receive feedback on performance accuracy as well as on intra-individual variability in reaction times. The software will be pilot tested in Phase I to determine performance thresholds and intervention duration. Also, focus groups will be conducted to obtain patient perceptions of each task's difficulty and interest level. In Phase II (R33 grant), a preliminary randomized clinical trial will be conducted in order to obtain initial estimates of treatment efficacy. Pre-, post-, and follow up outcomes will be collected on a wide range of neuropsychological, behavioral, and academic measures. Effect size estimates across outcomes will be used to guide sample size determinations for future clinical trials of multifaceted cognitive training.

ELIGIBILITY:
Inclusion Criteria:

* Consent: The family must provide signature of informed consent by parents or legal guardians.
* Age at time of Screening: 7 to 12 years of age, inclusive.
* Gender: includes male and female children.
* ADHD Diagnostic Status: ADHD patients must meet DSM-IV criteria for ADHD-PIT or ADHD-CT subtype. Section D.4 below describes in detail the diagnostic process for arriving at diagnosis.
* Cognitive Functioning: IQ of greater than 80 as estimated by the Wechsler Intelligence Scale for Children Fourth Edition.
* Learning Disability: Children must score 75 or above on two of the Wechsler Individual Achievement Test (WIAT) subtests (Reading & Numerical Operations).
* School: Children must be enrolled in a school setting from which teacher ratings can be obtained.
* History of Psychiatric Medications: Children may be taking psychiatric medications. However, they must present with significant ADHD inattention symptoms while on medication in order to be included in the study. We will ask that children on ADHD medications to refrain from altering the dosage for 10 weeks from study enrollment to after the immediate post-intervention follow-up. In order to screen for possible medication adjustments, all parents will be asked during the initial phone screen if their child is on an ADHD medication and if they anticipate a change in that medication dosage. If they answer that they anticipate a dosage change, they will be excluded from the study.

Exclusion Criteria:

* Understanding Level. The patient and parent cannot understand or follow instructions given in the study.
* Exclusionary Psychiatric Conditions: Children who meet diagnostic criteria on the K-SADS for OCD, any psychotic disorder, major depressive disorder or bipolar disorder will be excluded from participation.
* Developmental Disabilities. Patients will be excluded if they are deemed to be significantly developmentally delayed or have a pervasive developmental disorder. Developmental delay will be operationally defined as an IQ score below 80. Children scoring 80 or above will be included. A semi-structured interview, the CAARTE, will be used to screen for autism.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2011-04; Primary Completion 2013-12 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery N Epstein, Ph.D., Principal Investigator — Cincinnati Childrens Hospital Medical Center
Locations (1):
- Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Multifaceted Cognitive Training | Sham Cognitive Training
Started | 22 | 22
Completed | 17 | 18
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Multifaceted Cognitive Training | Sham Cognitive Training | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 22 | 44
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.05 (1.73) | 9.22 (1.65) | 9.14 (1.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 16 | 18 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 22 | 21 | 43
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 4 | 5
  White | 20 | 18 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Total ADHD Symptom Score From Vanderbilt ADHD Parent Rating Scale
Description: Total ADHD Symptom Score on the Parent Vanderbilt Rating Scales; range = 0-54; this score is computed by summing the 18 ADHD symptom items which are each rated on a 0-3 Likert scale (0="Never"; 1="Occasionally"; 2="Often"; 3="Very often"); higher scores indicate higher severity of ADHD symptoms.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Multifaceted Cognitive Training | Sham Cognitive Training
Number analyzed (Participants) | 17 | 18
units on a scale | 25.94 (8.95) | 28.28 (8.21)
Statistical Analysis 1: Comparison: Multifaceted Cognitive Training vs Sham Cognitive Training; Test type: Superiority or Other; p = .35, ANCOVA; Controlling for baseline scores

2. Secondary Outcome: Reaction Time Variability on go/No-go Task
Description: Standard deviation of reaction times for correct responses to Go trials on a Go/No-Go Task
Time Frame: 8 weeks
Population: Go/No-Go task data was not available for one participant in the Sham Cognitive Training condition
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Multifaceted Cognitive Training | Sham Cognitive Training
Number analyzed (Participants) | 17 | 17
milliseconds | 182.51 (96.12) | 160.25 (95.82)
Statistical Analysis 1: Comparison: Multifaceted Cognitive Training vs Sham Cognitive Training; Test type: Superiority or Other; p = .68, ANCOVA; Controlling for baseline scores

3. Secondary Outcome: Proportion of Words Read Accurately Using the AIMSWEB
Description: Number of words read correctly divided by number of words read
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: proportion of words read accurately
Arm/Group | Multifaceted Cognitive Training | Sham Cognitive Training
Number analyzed (Participants) | 17 | 18
proportion of words read accurately | .98 (.01) | .98 (.02)
Statistical Analysis 1: Comparison: Multifaceted Cognitive Training vs Sham Cognitive Training; Test type: Superiority or Other; p = .57, ANCOVA; Controlling for baseline scores

ADVERSE EVENTS:
Arm/Group | Multifaceted Cognitive Training | Sham Cognitive Training
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No